CLINICAL TRIAL: NCT04595539
Title: Does Attention Training Technique Enhance the Efficacy of Behavioral Activation Treatment for Depression: A Multiple Baseline Study
Brief Title: Intervention Targeting Depressive Symptoms and Mental Rumination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Audrey Krings, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1920-119
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-10

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Masking Description: A blinding procedure was used for the pre-post evaluations: interviews were recorded and each video or sound recording was evaluated at the end of the study by one (or two) independent evaluator who was unaware of the recordings' assessment time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simultaneous interventions (Experimental): In this condition, both interventions are proposed simultaneously. Condition 1 is spread over 5 weeks with 5 weekly laboratory sessions of 2-hours (one hour of BATD and one hour of ATT separated by a break). A 30-minutes ATT sessions at home were prescribed between sessions for a total of 5 laboratory ATT sessions and 5 at home ATT sessions.
  Interventions: Behavioral: Behavioral Activation treatment with Attention Training Technique
- Sequential interventions (Experimental): In this condition, the interventions are introduced sequentially. Condition 2 is spread over 7 weeks with 8 weekly laboratory sessions, 7 sessions of 1-hour and one session of 2-hours (Sessions 4 with of one hour of ATT followed by one hour of BATD separated by a break). A six 30-minutes ATT sessions were prescribed between the first 4 sessions of ATT for a total of 4 laboratory ATT sessions and 6 at home ATT sessions.
  Interventions: Behavioral: Behavioral Activation treatment with Attention Training Technique
- Sequential interventions in reverse order (Experimental): In this condition, the interventions are introduced sequentially in the reverse order than the condition 2. Condition 3 is spread over 7 weeks with 8 weekly laboratory sessions, 7 sessions of 1-hour and one session of 2-hours (Sessions 5 with of one hour of BATD followed by one hour of ATT separated by a break). A six 30-minutes ATT sessions were prescribed between the 4 last sessions for a total of 4 laboratory ATT sessions and 6 at home ATT sessions.
  Interventions: Behavioral: Behavioral Activation treatment with Attention Training Technique

INTERVENTIONS:
Behavioral: Behavioral Activation treatment with Attention Training Technique — The BATD includes the development of a shared formulation, psychoeducation, self-monitoring of daily activities, identifying "depressed behaviours", developing alternative goal orientated behaviours, scheduling of valued activities, and problem solving around difficulties implementing scheduled activities.
  Wells's Attention Training is a task designed to train selective attention to specific information by training individuals to attend to multiple auditory external sources. In addition to auditory exercices, the ATT sessions included psychoeducation, discussion around rumination (e.g. controllability, usefulness), self-report evaluation of self-focused before and after the auditory exercices, and transfer to everyday life.

SUMMARY:
This study aims to investigate the combine effects of Behavioral Activation and Attention Training on depression, well-being and other processes involved in depression as rumination.

A multiple baseline design is followed with multiple idiographic assessments, in addition to a pre-post and follow-up standardized assessment design.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is one of the most prevalent mental disorders, as well as one of the leading causes of disability worldwide. Behavioral activation is an empirically validated treatment for depression associated with medium effect size. The rationale of behavioral activation is to increase activation and reduce avoidance in order to reduce depressive affects. In parallel, Attention Training Techniques (ATT) is also an empirically validated treatment for depression. The rationale of ATT is to attenuate the self-focused attention and increase flexible attentional control over information processing to reduce depressive affects. ATT could target specific cognitive factors that are not changed through traditional interventions, and might enhance treatment outcomes for clinical and subclinical depressed when used in adjunct to psychotherapy. Then, the use of ATT may be a promising avenue to increase effectiveness of behavioral activation treatment.

The aims of the study are multiple. First, to measure the treatment feasibility and adherence of different treatment combinations and to measure it throughout the study. Second, to investigate the efficacy of Behavioral Activation Therapy for Depression combined with Attention Training sessions in subclinical and clinical depressed participants. Third, to investigate the mechanisms of change of both interventions.

The design will follow an "A1-B-A2'" design. Daily ideographic measures will be collected during all phases. Phase A1 and A2 are non-interventional phases of baseline and follow-up period respectively. Participants are randomly allocated to baseline lengths of 7, 10 and 15 days. Phase B is the intervention phase ranging from 5 weeks to 7 weeks. Three conditions exist with participants randomly allocated to one of these conditions. The intervention is provided in individual once a week. The first condition is a combination of 5 weeks of behavioral activation treatment for depression (BATD) and Attention Training technique (ATT)(2 hours/week). The second condition is 3 weeks of ATT followed by 5 weeks of BATD (1 hour/week), and the third is 5 weeks of BATD followed by 3 weeks of ATT (1 hour/week). Nomothetic standardized measures were also collected at pre-treatment (T0), after treatment (T1), after two weeks (T2) and 3 months later (T3).

The investigators hypothesized that the three proposed conditions will have an effect on the following target variables: activation, avoidance, reward motivation, self-focused attention, awareness as well as on transfer measures: depressive symptoms, rumination, anhedonia, well-being, social and work impairments, and cognitive control (2) changes in the target variables should preceded changes in the transfer measures (3) the therapeutic effects would be greater and faster when the treatments are combined than when they are offered sequentialy (i.e., in condition 1 versus conditions 2 and, (4) the therapeutic effect observed in Phase B was maintained in follow-up.

Target measures were expected to change with the introduction of intervention in comparison to baseline phase. In Condition of combination, the investigators expected to observe in Phase B an enhancement of activation, awareness and reward motivation and a decrease in avoidance and self-focused attention in comparison to the baseline phase. In Condition 2 with ATT sessions followed by BA sessions, the investigators expected to observe a reduction of self-focus attention, and an enhancement of awareness with the introduction of ATT, and an enhancement of activation and reward motivation and a reduction of avoidance with the introduction of BA. In Condition 3 with BA sessions followed by ATT sessions, the investigators expected the opposite pattern of change with first an enhancement of activation and reward motivation and a reduction of avoidance with the introduction of BA in comparison to baseline and then a reduction of self-focus attention, and an enhancement of awareness with the introduction of ATT in comparison to baseline.

ELIGIBILITY:
Inclusion Criteria:

* good understanding of French,
* at least a medium level of depressive symptoms
* report the presence of abstract rumination that generates negative mood.

Exclusion Criteria:

* Having a history of psychotic disorder
* Having a history of Bipolar disorder,
* Having a history of severe brain trauma or epilepsy
* with a moderate or severe substance use disorder other than tobacco (according to the DSM-V; i.e., showing 4 or more symptoms
* with an organic illness (e.g. cancer),
* with a concurrent additional psychotherapy,
* with acute suicidal ideation,
* with evidence of a significant change in medication within one month prior to baseline assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Depressive symptomatology | up to 72 hours before treatment
  The Beck depression inventory- second edition (BDI-II) is a 21-items scale that assesses the severity of depressive symptoms during the last two weeks. The score may range from 0 to 63. Higher score indicates higher depressive symptoms (worse outcome).
Depressive symptomatology | up to 72 hours after treatment
  The Beck depression inventory- second edition (BDI-II) is a 21-items scale that assesses the severity of depressive symptoms during the last two weeks.The score may range from 0 to 63. Higher score indicates higher depressive symptoms (worse outcome).
Depressive symptomatology | Two weeks after treatment
  The Beck depression inventory- second edition (BDI-II) is a 21-items scale that assesses the severity of depressive symptoms during the last two weeks.The score may range from 0 to 63. Higher score indicates higher depressive symptoms (worse outcome).
Depressive symptomatology | Three months after treatment
  The Beck depression inventory- second edition (BDI-II) is a 21-item scale that assesses the severity of depressive symptoms during the last two weeks.The score may range from 0 to 63. Higher score indicates higher depressive symptoms (worse outcome)
Activation | up to 72 hours before treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. Activation may range from 0 to 42. Higher scores indicate greater activation level (better outcome)
Activation | up to 72 hours after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. Activation may range from 0 to 42. Higher scores indicate greater activation level (better outcome).
Activation | Two weeks after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. Activation may range from 0 to 42. Higher scores indicate greater activation level (better outcome)
Activation | Three months after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. Activation may range from 0 to 42. Higher scores indicate greater activation level (better outcome)
Avoidance | up to 72 hours before treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. The score on behavioral avoidance may range from 0 to 30. Higher scores indicate greater behavioral avoidance (worse outcome).
Avoidance | up to 72 hours after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. The score on behavioral avoidance may range from 0 to 30. Higher scores indicate greater behavioral avoidance (worse outcome).
Avoidance | Two weeks after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. The score on behavioral avoidance may range from 0 to 30. Higher scores indicate greater behavioral avoidance (worse outcome).
Avoidance | Three months after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-item scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. The score on behavioral avoidance may range from 0 to 30. Higher scores indicate greater behavioral avoidance (worse outcome).
Social and Work Impairments | up to 72 hours before treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. The scores on Social and Work impairments may range from 0 to 30. Higher scores indicate higher Social and Work impairments respectively (worse outcomes)
Social and Work Impairments | up to 72 hours after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. The scores on Social and Work impairments may range from 0 to 30. Higher scores indicate higher Social and Work impairments respectively (worse outcomes)
Social and Work Impairments | Two weeks after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. The scores on Social and Work impairments may range from 0 to 30. Higher scores indicate higher Social and Work impairments respectively (worse outcomes)
Social and Work Impairments | Three months after treatment
  The Behavioral Activation for Depression Scale (BADS) is a 25-items scale that assesses behavioral activation. Five subscales have been identified: Activation, Behavioral Avoidance, Rumination, Work/School Impairment and Social Impairment. The scores on Social and Work impairments may range from 0 to 30. Higher scores indicate higher Social and Work impairments respectively (worse outcomes)
Mental Rumination | up to 72 hours before treatment
  The Revised version of Mini-CERTS (RTMQ) is a 18-items scale assessing repetitive thinking. Three subscales are identified, the first is characterized by thoughts at an abstract, overgeneral level that address the causes and consequences of one's mood or condition (named AERT). The second is characterized by a mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds (named CERTS). The third is characterized by a fluent and flexible thinking, with creative content (names CREATIVE). Higher scores indicate more abstract and general ruminative thinking for AERT (worse outcome), a more constructive way to ruminate for CERTS and CREATIVE (better outcome).
Mental Rumination | up to 72 hours after treatment
  The Revised version of Mini-CERTS (RTMQ) is a 18-items scale assessing repetitive thinking. Three subscales are identified, the first is characterized by thoughts at an abstract, overgeneral level that address the causes and consequences of one's mood or condition (named AERT). The second is characterized by a mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds (named CERTS). The third is characterized by a fluent and flexible thinking, with creative content (names CREATIVE). Higher scores indicate more abstract and general ruminative thinking for AERT (worse outcome), a more constructive way to ruminate for CERTS and CREATIVE (better outcome).
Mental Rumination | Two weeks after treatment
  The Revised version of Mini-CERTS (RTMQ) is a 18-items scale assessing repetitive thinking. Three subscales are identified, the first is characterized by thoughts at an abstract, overgeneral level that address the causes and consequences of one's mood or condition (named AERT). The second is characterized by a mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds (named CERTS). The third is characterized by a fluent and flexible thinking, with creative content (names CREATIVE). Higher scores indicate more abstract and general ruminative thinking for AERT (worse outcome), a more constructive way to ruminate for CERTS and CREATIVE (better outcome).
Mental Rumination | Three months after treatment
  The Revised version of Mini-CERTS (RTMQ) is a 18-items scale assessing repetitive thinking. Three subscales are identified, the first is characterized by thoughts at an abstract, overgeneral level that address the causes and consequences of one's mood or condition (named AERT). The second is characterized by a mode of thinking centered on how one is presently feeling and experiencing the ongoing situation, and how a present experience unfolds (named CERTS). The third is characterized by a fluent and flexible thinking, with creative content (names CREATIVE). Higher scores indicate more abstract and general ruminative thinking for AERT (worse outcome), a more constructive way to ruminate for CERTS and CREATIVE (better outcome).
Well-being | up to 72 hours before treatment
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-items scale assessing mental well-being. The score may range from 14 to 70. Higher scores indicate higher mental well-being (better outcome).
Well-being | up to 72 hours after treatment
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-items scale assessing mental well-being. The score may range from 14 to 70. Higher scores indicate higher mental well-being (better outcome).
Well-being | Two weeks after treatment
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-items scale assessing mental well-being. The score may range from 14 to 70. Higher scores indicate higher mental well-being (better outcome).
Well-being | Three months after treatment
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a 14-items scale assessing mental well-being. The score may range from 14 to 70. Higher scores indicate higher mental well-being (better outcome).
Anhedonia | up to 72 hours before treatment
  The Savoring belief Inventory (SBI) is an 24-items scale assessing individuals' attitudes regarding savoring positive experiences. Three subscales related to three temporal orientations are identified, one related to the past (reminiscence), one related to the present moment (present), and one related to the future (anticipation) each represented by 8 items. Higher scores indicate higher level of approach and savor pleasant events (better outcome).
Anhedonia | up to 72 hours after treatment
  The Savoring belief Inventory (SBI) is an 24-items scale assessing individuals' attitudes regarding savoring positive experiences. Three subscales related to three temporal orientations are identified, one related to the past (reminiscence), one related to the present moment (present), and one related to the future (anticipation) each represented by 8 items. Higher scores indicate higher level of approach and savor pleasant events (better outcome).
Anhedonia | Two weeks after treatment
  The Savoring belief Inventory (SBI) is an 24-items scale assessing individuals' attitudes regarding savoring positive experiences. Three subscales related to three temporal orientations are identified, one related to the past (reminiscence), one related to the present moment (present), and one related to the future (anticipation) each represented by 8 items. Higher scores indicate higher level of approach and savor pleasant events (better outcome).
Anhedonia | Three months after treatment
  The Savoring belief Inventory (SBI) is an 24-items scale assessing individuals' attitudes regarding savoring positive experiences. Three subscales related to three temporal orientations are identified, one related to the past (reminiscence), one related to the present moment (present), and one related to the future (anticipation) each represented by 8 items. Higher scores indicate higher level of approach and savor pleasant events (better outcome).
Cognitive control. | up to 72 hours before treatment
  A computerized version of the Paced Auditory Serial- Addition Task was used as a measure of participants' updating abilities reflecting the working memory ability (PASAT). Higher scores suggest greater cognitive control ressources (better outcome).
Cognitive control. | up to 72 hours after treatment
  A computerized version of the Paced Auditory Serial- Addition Task was used as a measure of participants' updating abilities reflecting the working memory ability (PASAT). Higher scores suggest greater cognitive control ressources (better outcome).
Cognitive control. | Two weeks after treatment
  A computerized version of the Paced Auditory Serial- Addition Task was used as a measure of participants' updating abilities reflecting the working memory ability (PASAT). Higher scores suggest greater cognitive control ressources (better outcome).
Cognitive control. | Three months after treatment
  A computerized version of the Paced Auditory Serial- Addition Task was used as a measure of participants' updating abilities reflecting the working memory ability (PASAT). Higher scores suggest greater cognitive control ressources (better outcome).
Attention Style Questionnaire | up to 72 hours before treatment
  The Attentional Style Questionnaire (ASQ) is a 12- items scale assessing the capacity of an individual to maintain attention on task-related stimuli and not to be distracted by interfering stimuli. Two factors are identified: externally and internally oriented attention. Higher score indicating a marked bottom-up oriented attentional style, and a lower score indicating a marked top-down oriented attentional style.
Attention Style Questionnaire | up to 72 hours after treatment
  The Attentional Style Questionnaire (ASQ) is a 12- items scale assessing the capacity of an individual to maintain attention on task-related stimuli and not to be distracted by interfering stimuli. Two factors are identified: externally and internally oriented attention. Higher score indicating a marked bottom-up oriented attentional style, and a lower score indicating a marked top-down oriented attentional style.
Attention Style Questionnaire | Two weeks after treatment
  The Attentional Style Questionnaire (ASQ) is a 12- items scale assessing the capacity of an individual to maintain attention on task-related stimuli and not to be distracted by interfering stimuli. Two factors are identified: externally and internally oriented attention. Higher score indicating a marked bottom-up oriented attentional style, and a lower score indicating a marked top-down oriented attentional style.
Attention Style Questionnaire | Three months after treatment
  The Attentional Style Questionnaire (ASQ) is a 12- items scale assessing the capacity of an individual to maintain attention on task-related stimuli and not to be distracted by interfering stimuli. Two factors are identified: externally and internally oriented attention. Higher score indicating a marked bottom-up oriented attentional style, and a lower score indicating a marked top-down oriented attentional style.

SECONDARY OUTCOMES:
Multiple measures of Activation | everyday through study completion (an average of 7 to 9 weeks)
  Activation level was collected daily at the end of the day in a booklet with the following item "I have been an active person and have accomplished the goals I set for myself." accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely).
Multiple measures of reward motivation | everyday through study completion (an average of 7 to 9 weeks)
  Reward motivation was collected daily at the end of the day in a booklet with the following item "I am looking forward to some upcoming events or activities" accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely).
Multiple measures of Avoidance | everyday through study completion (an average of 7 to 9 weeks)
  Avoidance was collected daily at the end of the day in a booklet with the following item "Most of what I did was to escape from or avoid something unpleasant." accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely).
Multiple measures of focus of attention | everyday through study completion (an average of 7 to 9 weeks)
  Focus of attention was collected daily at the end of the day in a booklet with the following item "I focused my attention on myself rather than on my external environment." accompanied by a Visual Analogue Scale (ranging from left side : not at all to right side completely).
Multiple measures of awareness | everyday through study completion (an average of 7 to 9 weeks)
  Awareness was collected daily at the end of the day in a booklet with the following item "I was aware of my thoughts, body sensations, emotions and feelings" accompanied by a Visual Analogue Scale (ranging from left side : not at all to right side completely).
Multiple measures of Rumination | everyday through study completion (an average of 7 to 9 weeks)
  Rumination was collected daily at the end of the day in a booklet with the following item ". I spent a long time thinking over and over about my problems." accompanied by a Visual Analogue Scale (ranging from left side : not at all to right side completely).
Multiple individual measures of depressive symptoms | everyday through study completion (an average of 7 to 9 weeks)
  Two items assessing depressive symptoms were selected by the participant based on a idiographic approach. For exemple : "I had difficulty to experience pleasure in what I did", "I felt tired", "I felt like I was being punished", "I had a hard time getting interested in anything", "I've been irritable", "I felt guilty", "I felt sad". Depressive symptoms were collected at the end of the day in a booklet with two items accompanied by Visual Analogue Scales (ranging from left side : not at all to right side completely).
Multiple individual measures of functioning on disturbed area of life | everyday through study completion (an average of 7 to 9 weeks)
  Two items assessing disturbed functioning on area of life (e.g. social, professional, daily skills, hobbies, family, or relationships) were selected by the participant based on a idiographic approach. Depressive symptoms were collected at the end of the day in a booklet with two items accompanied by Visual Analogue Scales (ranging from left side : not at all to right side completely).
Multiple individual measures of personal complaints not related to the intervention. | everyday through study completion (an average of 7 to 9 weeks)
  One item assessing personal complaints (e.g. impulsivity, assertiveness, sleep) was selected by the participant based on a idiographic approach. Personal complaints was collected at the end of the day in a booklet with two items accompanied by Visual Analogue Scales (ranging from left side : not at all to right side completely).
Multiple measures of mood | everyday through study completion (an average of 7 to 9 weeks)
  Mood was collected daily at the end of the day in a booklet with items accompanied by a Visual Analogue Scale (ranging from left side : very negative to right side very positive).
Credibility and Expectancy | Up to 72 hours after the beginning of interventions and through intervention completion (an average of 5 to 7 weeks).
  The Credibility and expectancy of treatment Questionnaire (CEQ) is a 6-items scale that assesses the therapy credibility who refers to the extent to which a treatment makes sense, is believable, convincing and logical, and the expectancy who refers to improvements that patients believe will occur with the intervention. Two subscales are identified: the Credibility and the Expectancy. Higher scores indicate better credibility and Expectancy from the patients (better outcome).
Therapeutic alliance | Up to 72 hours after the beginning of interventions and through intervention completion (an average of 5 to 7 weeks).
  The Helping Alliance Questionnaire (HAQ) is a 8-items scale that assesses client-reported quality of the therapeutic alliance. Higher score indicated higher client satisfaction in the therapeutic alliance (better outcome).
Client Satisfaction | up to 72 hours after treatment
  The Consumer Satisfaction Questionnaire (CSQ) is a 8-items scale that assesses client satisfaction with treatment. Higher score indicates greater satisfaction.
Client adherence and satisfaction | up to 72 hours after treatment
  This post intervention interview focused on satisfaction with the organization (i.e., size of the group, rhythm of progression, materials given, sessions' length, sessions' frequency, location, equipment), with the content (i.e., pertinence to everyday life, helpfulness of tools and compatibility with their expectations, identification, applicability, improvement, feedback) and with the therapists (i.e., motivation, communication skills, knowledge, adaptation abilities).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Blairy, Study Director — University of Liege
Locations (1):
- Liège University, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No
Data and analyses will be available from an online repository or from the principal investigator